CLINICAL TRIAL: NCT03596034
Title: A Study to Characterize Puff Topography With Use of a JUUL 5% Electronic Nicotine Delivery Systems (ENDS) in Adult Smokers
Brief Title: A Study to Characterize Puff Topography With Use of JUUL 5% Electronic Nicotine Delivery Systems (ENDS) in Adult Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Juul Labs, Inc. (Industry)
Collaborators: Rose Research Center, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Protocol No.755-00042
Record Dates: First submitted 2018-06-06; First posted 2018-07-23 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2018-10

CONDITIONS: Tobacco Use; Nicotine Dependence, Other Tobacco Product; Tobacco Smoking
Keywords: Electronic Nicotine Delivery System (ENDS); ENDS; Puff Topography
MeSH Terms: conditions — Tobacco Use; Tobacco Use Disorder; Tobacco Smoking; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- JUUL 5%, Virginia Tobacco, ENDS product (Experimental): Subjects participate in a 15 day product use period during which subjects will be requested to predominantly use the JUUL 5% product ad libitum as their primary source of nicotine. Subjects will be asked to report their daily use of the JUUL 5% product and combustibles per day (CPD) throughout the 15 day product use period.
  Interventions: Other: JUUL 5%, Virginia Tobacco, ENDS product

INTERVENTIONS:
Other: JUUL 5%, Virginia Tobacco, ENDS product — Subjects participate in a 15 day product use period during which subjects will be requested to predominantly use the JUUL 5% product ad libitum as their primary source of nicotine. Subjects will be asked to report their daily use of the JUUL 5% product and CPD throughout the 15 day product use period.
  Other Names: ENDS

SUMMARY:
A Study to Characterize Puff Topography with Use of a JUUL 5% Electronic Nicotine Delivery Systems (ENDS) in Adult Smokers

DETAILED DESCRIPTION:
This will be an open label study to evaluate puff topography in adult smokers using a JUUL 5% ENDS. Up to 30 subjects will be enrolled and evaluated on Day 1 and Day 15. The duration of the study is 15 days with up to a 28 days screening window.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy, adult, male or female smoker, 21 to 65 years of age
2. Has been a smoker for at least 12 months prior to Screening.
3. Currently smokes an average of 5 to 40 manufactured combustible (menthol or non menthol) cigarettes per day.
4. A female subject of childbearing potential must have been using 1 of the following forms of contraception and agree to continue using it through completion of the study
5. Provides voluntary consent to participate in this study documented on the signed informed consent form.

Key Exclusion Criteria:

1. Has a clinically significant abnormal finding on the physical examination, medical history, vital signs, ECG, or clinical laboratory results, in the opinion of the PI.
2. Has a body mass index (BMI) > 40 kg/m2 or < 18 kg/m2 at Screening.
3. Has a history of drug or alcohol abuse within 24 months of Day 1.
4. If female, the subject is pregnant, lactating, or intends to become pregnant during the time period from Screening through the end of study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Puff Topography Parameter - Puff Duration | 15 days
  To characterize overall puff duration
Puff Topography Parameter - Puff Volume | 15 days
  To characterize overall puff volume
Puff Topography Parameter - Peak Puff Flow Rate | 15 days
  To characterize overall peak puff flow rate
Puff Topography Parameter - Average Puff Flow Rate | 15 days
  To characterize overall average puff flow
Puff Topography Parameter - Inter-Puff Interval | 15 days
  To characterize overall inter-puff interval (time between puffs)

SECONDARY OUTCOMES:
Self-reported product use over 15-day period | 15 days
  To assess the relationship between puff topography parameters and self-reported product use (number of puffs per day and number of JUULpods started each day) in a 15-day product use period.
Subjective measure of product liking | 15 days
  To assess the relationship between puff topography parameters and JUUL 5% ENDs liking using a "Product Liking Questionnaire". Visual analogue scale with scale 0 (Not at all) to 100 (Extremely) in response to question "I like using the JUUL Product."
Subjective measure of cigarette dependence | 15 days
  Assessment of cigarette dependence with "Fagerstrom Test for Cigarette Dependence Questionnaire (FTCD)". Questionnaire consists of 6 questions.
Subjective measure of smoking urges | 15 days
  Assessment of current smoking urge with "Questionnaire of Smoking Urges - Brief (QAU-B)". Responses to various statements with scale 1 (Strongly Disagree) to 7 (Strongly Agree).
Subjective measure of effects of nicotine | 15 days
  Assessment of nicotine using the "Direct Effects of Nicotine Scale." Visual analogue scale with scale 0 (Not at All) to 100 (Extremely) in response to words describing how the subject feels.
Subject measure of affect | 15 days
  Assessment of affect using the "Positive and Negative Affect Scale (PANAS)". Scale consists of a number of words that describe different feelings and emotions. Scale 1 (Very Slightly or Not at All), 2 (A Little), 3 (Moderately), 4 (Quite a Bit), 5 (Extremely).
Subjective measure of nicotine withdrawal | 15 days
  Assessment of nicotine withdrawal using the "Nicotine Withdrawal Scale (MNWS-R)." Scale consists of 15 words/statements that describe different feelings. Scale 0 (None) to 4 (Severe).

CONTACTS AND LOCATIONS:
Overall Officials: Jed Rose, MD, Principal Investigator — Rose Research Center, LLC
Locations (2):
- United States (2):
  - Rose Research Center Charlotte, Charlotte, North Carolina
  - Rose Research Center Raleigh, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided